CLINICAL TRIAL: NCT00296907
Title: Psychological Interventions in Siblings of Children With Cancer: a Randomized Controlled Study
Brief Title: Psychological Interventions in Siblings of Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PIGO-1
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Cancer
Keywords: cancer; siblings; behavior; psychological adaptation; intervention
MeSH Terms: conditions — Neoplasms; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Psychological Intervention (Experimental): 2-session psychological intervention
  Interventions: Behavioral: Brief psychological intervention

INTERVENTIONS:
Behavioral: Brief psychological intervention — Psychoeducation, provision of medical knowledge, coping skills training

SUMMARY:
The purpose of the study is to evaluate the effectiveness of a two-session brief psychological intervention in siblings of pediatric cancer patients with regard to behavior problems and depression.

DETAILED DESCRIPTION:
Within a randomized controlled design the effects of a brief two-session psychological intervention (child, parents) shall be studied in 30 siblings of newly diagnosed pediatric cancer patients. After a baseline assessment 3-4 weeks after diagnosis participants are randomly assigned to an intervention or waiting list group. Both are re-assessed at 3 and 6 months by means of standardized questionnaires assessing psychological adaptation and behavior. The intervention is provided to the waiting list group after the 6-month assessment.

ELIGIBILITY:
Inclusion Criteria:

brother or sister with newly diagnosed cancer treated at the University Children's Hospital command of the German language normal developmental level

Exclusion Criteria:

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
KIDSCREEN: health-related quality of life | baseline, 3 and 6 months post intervention
UCLA Child PTSD Reaction Index | baseline, 3 and 6 months post intervention
DIKJ (Depression-Inventory for Children and Adolescents) | baseline, 3 and 6 months post intervention
Child Behavior Checklist | Baseline, 3 and 6 months post intervention
Spence Children's Anxiety Scale | baseline, 3 and 6 months post intervention

SECONDARY OUTCOMES:
Posttraumatic Distress Scale | baseline, 3 and 6 months post intervention
Symptom Checklist 27 | baseline, 3 and 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Landolt, PhD, Principal Investigator — University Children's Hospital Zurich, Psychosomatic and Psychiatry
Locations (1):
- University Children's Hospital Zurich, Psychosomatic and Psychiatry, Zurich, Switzerland

REFERENCES:
- [Result] Prchal A, Graf A, Bergstraesser E, Landolt MA. A two-session psychological intervention for siblings of pediatric cancer patients: a randomized controlled pilot trial. Child Adolesc Psychiatry Ment Health. 2012 Jan 11;6(1):3. doi: 10.1186/1753-2000-6-3. PMID 22236392